CLINICAL TRIAL: NCT07236788
Title: Study on Supplement of Intravenous Ferric Derisomaltose to Prevent Anemia and Improve the Quality of Life in Obese Patients With Iron Deficiency.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Director of the General Surgery Department & Obesity and Metabolic Disease Center of China-Japan Friendship Hospital, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-HX-133
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Anemia; Iron Deficiencies; Bariatric Surgery
MeSH Terms: conditions — Obesity; Anemia; Iron Deficiencies | interventions — iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 3±1 days before the operation, intravenous infusion of isomaltose iron injection was administered. The dosage was in accordance with the drug instructions. The maximum single infusion dose was 20mg/kg. If the dose could not be made up in one infusion, the remaining dose should be made up every other week.
  Interventions: Drug: Iron Isomaltoside injection
- Placebo group (Placebo Comparator): At the same time point, the same dose of physiological saline was infused.
  Interventions: Drug: Physiological saline solution (as placebo)

INTERVENTIONS:
Drug: Iron Isomaltoside injection — Patients in the isomaltan iron group received intravenous isomaltan iron dissolved in 250 ml of normal saline 3 days prior to surgery. The patients' iron requirements were calculated using a simplified scale, with a maximum single dose of 20 mg/kg. If the dose was insufficient in a single administration, a second infusion was required every other week. The placebo group received an equal volume of 0.9% normal saline.
  Simplified scale:
  Hemoglobin (g/L) patient weight <50kg 50-70kg >70kg
  ≥100 500mg 1000mg 1500mg <100 500mg 1500mg 2000mg
  Arms: Treatment group
Drug: Physiological saline solution (as placebo) — At the same time point, the same dose of physiological saline was infused as the experimental group.
  Arms: Placebo group

SUMMARY:
This study aimed to explore the effects of preoperative intravenous isomaltose iron supplementation versus placebo on postoperative Hb improvement, prevention of postoperative anemia, and improvement in quality of life in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* ① Baseline Hb: Men 10-14 g/dL, Women 10-13 g/dL; ② Iron deficiency: Serum ferritin (SF) <100 μg/L, and transferrin saturation (TSAT) <20%; ③ BMI >30 kg/m2.

Exclusion Criteria:

* ① Known severe hypersensitivity reactions to other parenteral iron supplements; ② Mean corpuscular volume (MCV) > 100 fL; ③ Received intravenous iron infusion within the past 3 months; ④ Concurrent tumors; ⑤ Concurrent iron overload or other hematologic disorders; ⑥ Concurrent infectious diseases such as hepatitis B; ⑦ Moderately impaired liver function: decompensated cirrhosis or hepatitis, ALT, AST > 3 × upper limit of normal (ULN); ⑧ Concurrent acute or chronic infections, heart failure, or other diseases affecting iron metabolism; ⑨ Patients with stage 3 or higher chronic renal insufficiency: glomerular filtration rate (eGFR) < 60 ml/min; ⑩ Pregnant or lactating women; ⑪ Acute infections, rheumatoid arthritis, or significant joint inflammation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
changes in Hb concentration compared to baseline | 3 months post-surgery,

SECONDARY OUTCOMES:
Incidence of anemia | 3 months, 6 months and 12 months after surgery
Iron metabolism indicators (serum ferritin, serum iron, total iron binding capacity, transferrin saturation) | 3 months, 6 months, and 12 months post-surgery
The proportion of patients requiring re-treatment for iron deficiency anemia within 12 months post-surgery (Hb < 11 g/dL, SF < 30 μg/L, or SF < 100 μg/L and TSAT < 20%). | 12 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China